CLINICAL TRIAL: NCT05524649
Title: Safety, Tolerability and Effect on Fecal Microbiota Composition of Two Probiotic Strains in Infants
Brief Title: Effect of Probiotics on Infant's Fecal Microbiota Composition
Acronym: BABYCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AB-BABYCARE-21
Record Dates: First submitted 2022-08-26; First posted 2022-09-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Microbial Colonization
Keywords: Probiotics; Infants; Microbiota
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled trial in 120 healthy infants between 1 and 90 days of age, who will be allocated to receive either one of the probiotic strains or placebo for 3 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Every product will be provided in identical packaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental 1 (Experimental): Probiotic single strain formulation comprising Bifidobacterium longum CECT7894 in liquid format suspended in sunflower oil. This probiotic strain has Qualified Presumption of Safety (QPS) status by European Food Safety Authority.
  Interventions: Dietary Supplement: Food Supplement 1
- Experimental 2 (Experimental): Probiotic single strain formulation comprising Pediococcus pentosaceus CECT8330 in liquid format suspended in sunflower oil. This probiotic strain has Qualified Presumption of Safety (QPS) status by European Food Safety Authority.
  Interventions: Dietary Supplement: Food Supplement 2
- Placebo (Placebo Comparator): Sunflower oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Food Supplement 1 — Probiotic single strain formulation containing Bifidobacterium longum CECT7894 for 3 months 5 drops/day
  Arms: Experimental 1
Dietary Supplement: Food Supplement 2 — Probiotic single strain formulation containing Pediococcus pentosaceus CECT8330 for 3 months 5 drops/day
  Arms: Experimental 2
Dietary Supplement: Placebo — 5 drops/day for 3 months of sunflower oil
  Arms: Placebo

SUMMARY:
Randomized clinical trial to evaluate the effect of two probiotic strains which belong to Bifidobacterium Longum and Pediococcus pentosaceus species on fecal microbiota composition in healthy infants. Secondary outcomes comprise evaluation of anthropometric growth, digestive tolerance, sleeping habits, incidence of functional gastrointestinal disorders, incidence of gastrointestinal and respiratory infections, allergic reactions and safety and tolerability of the product.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled clinical trial to determine the effect of the probiotic strains Bifidobacterium longum and Pediococcus pentosaceus on fecal microbiota composition in infants. Healthy babies with ages comprised between 60 and 90 days who meet inclusion and exclusion criteria will be randomized 1:1:1 to one of the following study groups: one group will receive Bifidobacterium longum, another group will receive Pediococcus pentosaceus and the other one will receive placebo for 3 months. Other study outcomes comprise anthropometric growth, frequency and consistency of the stools, digestive tolerance, wellbeing, number, type and duration of infections and functional gastrointestinal disorders, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants
* Age between 1 and 90 days
* Gestational age between 37 and 42 weeks
* Appropiate birth weight for gestational age (between P10 and P90)
* APGAR test score for birth normal at 1' and 5' of 7-10
* Whose parents accept the follow-up of the study procedures and sign the informed consent

Exclusion Criteria:

* Infants participating in other clinical study
* Fed with infant formula containing probiotics or other aliments or food supplement based in probiotics 4 weeks prior the start of the study
* Infants who have taken antibiotics 4 weeks prior the start study
* Infants with cow's milk protein allergy, lactose intolerance or other digestive diseases
* Mother's pathological background and during gestation: neurologic disorders, matabolopaties, diabetes mellitus type 1, chronic disease (hypothyroidism), maternal malnutrition
* Acute congenital or acquired diseases which can interfere with the growth and the normal feeding of the infant
* TORCH complex infections
* Every other diseases related with the immune system
* Parents who can not accomplish the follow-up of the study (medical criterium)

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Bifidobacterium longum and Pediococcus pentosaceus in feces | day 0, month 3
  Change of total counts of Bifidobacterium longum and Pediococcus pentosaceus in feces determined by qPCR

SECONDARY OUTCOMES:
Weight change | day 0, month 1, month 2, month 3
  Change in weight (g per day) between day 0 and month 3
Length change | day 0, month 1, month 2, month 3
  Change in length (cm) between day 0 and month 3
Head circumference change | day 0, month 1, month 2, month 3
  Change in head circumference (cm) between day 0 and month 3
BMI change | day 0, month 1, month 2, month 3
  Change in BMI (kg/m2) between day 0 and month 3
Frequency of depositions | day 0, month 1, month 2, month 3
  Frequency of depositions (number stools/day) documented in participants diary
Consistency of stools | day 0, month 1, month 2, month 3
  Consistency of stools through a 5-item scale: 1= hard balls, 2=hard-formed, 3=soft-formed, 4=half liquid and 5=liquid
Infant colic | day 0, month 1, month 2, month 3
  Incidence of infant colic, defined as prolonged and recurrent periods of crying, agitation, or irritability without apparent cause that cannot be prevented or resolved by your caregivers, for three or more hours daily for three or more days a week
Vomiting | day 0, month 1, month 2, month 3
  Incidence of vomiting (n/day)
Sleeping habits | day 0, month 1, month 2, month 3
  Nocturnal sleeping (min/day), total sleeping hours (min/day)
Incidence of infections | day 0, month 1, month 2, month 3
  Number and duration (in days) of any type of infectious episodes
Fever | day 0, month 1, month 2, month 3
  Number of days with fever (axial body temperature higher than 37.5 ºC)
Antibiotics | day 0, month 1, month 2, month 3
  Number of days with antibiotic treatment
Change in fecal microbiota composition | day 0, month 3
  Analysis of α y β biodiversity, relative abundance of bacteria determined by 16S sequencing
sIgA in stool samples | day 0, month 3
  Analysis of secretory Immunoglobulin A (sIgA) in stools through ELISA
Calprotectin | day 0, month 3
  Analysis of fecal calprotectin through ELISA

CONTACTS AND LOCATIONS:
Locations (2):
- Instituto Nacional de Pediatría Insurgentes Sur 3700-C, Insurgentes Cuicuilco, Alcaldía Coyoacán, Puebla, Mexico
- Clínica Viamed Montecanal, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen K, Liu C, Li H, Lei Y, Zeng C, Xu S, Li J, Savino F. Infantile Colic Treated With Bifidobacterium longum CECT7894 and Pediococcus pentosaceus CECT8330: A Randomized, Double-Blind, Placebo-Controlled Trial. Front Pediatr. 2021 Sep 10;9:635176. doi: 10.3389/fped.2021.635176. eCollection 2021. PMID 34568236
- [Background] Braegger C, Chmielewska A, Decsi T, Kolacek S, Mihatsch W, Moreno L, Piescik M, Puntis J, Shamir R, Szajewska H, Turck D, van Goudoever J; ESPGHAN Committee on Nutrition. Supplementation of infant formula with probiotics and/or prebiotics: a systematic review and comment by the ESPGHAN committee on nutrition. J Pediatr Gastroenterol Nutr. 2011 Feb;52(2):238-50. doi: 10.1097/MPG.0b013e3181fb9e80. PMID 21150647
- [Background] Castanet M, Costalos C, Haiden N, Hascoet JM, Berger B, Sprenger N, Grathwohl D, Brussow H, De Groot N, Steenhout P, Pecquet S, Benyacoub J, Picaud JC. Early Effect of Supplemented Infant Formulae on Intestinal Biomarkers and Microbiota: A Randomized Clinical Trial. Nutrients. 2020 May 20;12(5):1481. doi: 10.3390/nu12051481. PMID 32443684
- [Background] Hoy-Schulz YE, Jannat K, Roberts T, Zaidi SH, Unicomb L, Luby S, Parsonnet J. Safety and acceptability of Lactobacillus reuteri DSM 17938 and Bifidobacterium longum subspecies infantis 35624 in Bangladeshi infants: a phase I randomized clinical trial. BMC Complement Altern Med. 2016 Feb 2;16:44. doi: 10.1186/s12906-016-1016-1. PMID 26832746
- [Background] Navarro-Tapia E, Sebastiani G, Sailer S, Toledano LA, Serra-Delgado M, Garcia-Algar O, Andreu-Fernandez V. Probiotic Supplementation During the Perinatal and Infant Period: Effects on Gut Dysbiosis and Disease. Nutrients. 2020 Jul 27;12(8):2243. doi: 10.3390/nu12082243. PMID 32727119
- [Background] Radke M, Picaud JC, Loui A, Cambonie G, Faas D, Lafeber HN, de Groot N, Pecquet SS, Steenhout PG, Hascoet JM. Starter formula enriched in prebiotics and probiotics ensures normal growth of infants and promotes gut health: a randomized clinical trial. Pediatr Res. 2017 Apr;81(4):622-631. doi: 10.1038/pr.2016.270. Epub 2016 Dec 21. PMID 28002391